<u>ID3 Medical - 20211119</u> BELSTREAM - Bard

## NCT03349996 Unique Protocol ID: ID3-20170704

## PROTOCOL SYNOPSIS: BELSTREAM study

| Title | Belgian Physician-Initiated Trial Investigating the Lifestream Peripheral Stent Graft System for the treatment of complex TASC C and D iliac lesions | |
|---|---|---|
| Objective | The objective of this clinical investigation is to evaluate, in a controlled setting, the | |
| | long-term (up to 60 months) safety and efficacy of the Lifestream Peripheral Stent | |
| | Graft System (Bard) in clinical settings post CE-certification when used according to | |
| | the indications of the IFU. | |
| Methodology | Prospective, multi-center, physician-sponsored clinical study | |
| Enrollment | 70 subjects | |
| Primary Endpoint | Efficacy | The primary endpoint of the study is primary patency at 12 months , |
| | endpoint | defined as a target lesion without a hemodynamically significant |
| | | stenosis on duplex ultrasound (>50%, systolic velocity ratio greater than |
| | | 2.5) and with freedom from Target Lesion Revascularization (TLR) within |
| | | 12 months. TLR is defined as a repeated intervention to maintain or re- |
| | | establish patency within the region of the treated arterial vessel plus |
| | | 5mm proximal and distal to the treated lesion edge. |
| | Safety | The primary safety endpoint of the study is the freedom of |
| | endpoint | periprocedural Serious Adverse Events (SAEs), defined according to ISO |
| | Ciraponit | 14155:2011 as any clinical event that is fatal, life-threatening, or judged |
| | | to be severe by the investigator; resulted in persistent or significant |
| | | disability; necessitated surgical or percutaneous intervention; or |
| | | required prolonged hospitalization. |
| Secondary Endpoint | 1. | Primary patency rate at 1-, 6-, 24-, 36-, 48- and 60 month follow-up. |
| | | Patients that present without a hemodynamically significant stenosis at |
| | | the target area on duplex ultrasound (>50%, systolic velocity ratio |
| | | greater than 2.5) and without prior TLR are defined as being primary |
| | | patent at the given follow-up. |
| | 2. | Stent graft occlusion rate at pre-discharge, 1-, 6-, 12-, 24-, 36-, 48-, and |
| | | 60-month follow-up. |
| | 3. | Ankle Brachial Index (ABI) at 1-, 6-, 12-, 24-, 36-, 48- and 60 month follow- |
| | | up compared with the baseline ABI. |
| | 4. | Amputation rate at 1-, 6-, 12-, 24-, 36-, 48- and 60 month follow-up, |
| | | defined as any amputation above the knee. |
| | 5. | Technical success, defined as the ability to achieve final residual |
| | | angiographic stenosis no greater than 30%. |
| | 6. | Clinical success at follow-up is defined as an improvement of Rutherford |
| | | classification at 1-, 6-, 12-, 24-, 36-, 48- and 60 -month follow-up of one |
| | | class or more as compared to the pre-procedure Rutherford |
| | | classification. |
| Inclusion Criteria | General inclusion criteria | |
| | 1. | Corresponding to the CE-mark indications/contra-indications and |
| | | according to the current medical guidelines for minimally invasive |
| | | peripheral interventions. |
| | 2. | Patient presenting with a stenotic or occlusive lesion at the iliac arteries |
| | | suitable for stenting (on indication for primary stenting, based on the |
| | 2 | discretion of the investigator) |
| | 3. | Patient presenting a score from 2 to 4 following Rutherford classification |
| | 4. | Patient is willing to comply with specified follow-up evaluations at the |
| | _ | specified times for the duration of the study |
| | 5. | Patient is >18 years old |

V2.00 dd20211119 1/4

<u>ID3 Medical - 20211119</u> BELSTREAM - Bard

| | 6. | Patient (or their legal representative) understands the nature of the |
|---|---|---|
| | 0. | procedure and provides written informed consent, prior to enrolment in |
| | | the study |
| | 7. | Patient is eligible for treatment with the Lifestream Peripheral Stent Graft |
| | | System (Bard) |
| | | raphic inclusion criteria |
| | 1. | The target lesion is either a modified TASC-II class C or D lesion with one of the listed specifications: |
| | | Type C lesions |
| | | Bilateral Common Iliac Artery occlusions |
| | | Bilateral External Iliac Artery stenoses 3–10 cm |
| | | long not extending into the Common Femoral |
| | | Artery |
| | | <ul> <li>Type D lesions</li> </ul> |
| | | <ul> <li>Unilateral occlusions of both Common Iliac</li> </ul> |
| | | and External Iliac Artery |
| | | <ul> <li>Diffuse disease involving the aorta bifurcation</li> </ul> |
| | | Bilateral occlusions of External Iliac Artery |
| | 2. | The target lesion has angiographic evidence of stenosis or restenosis post |
| | | PTA >50% or occlusion which can be passed with standard guidewire |
| | 3. | manipulation There is angiographic evidence of a patent Common and Deep Femoral |
| | ٥. | Artery |
| Exclusion criteria | 1. | PTA is technically not possible (not feasible to access the lesion or a |
| | | defect with the guidewire or balloon catheter) |
| | 2. | Presence of an aneurysm immediately adjacent to the site of stent graft |
| | | implantation |
| | 3. | Lesions in or adjacent to essential collaterals(s) |
| | 4. | Lesions in locations subject to external compression |
| | 5. | Heavily calcified lesions resistant to PTA |
| | 6.<br>7. | Patients with a history of secondation disorders |
| | 8. | Patients with a history of coagulation disorders Patients with aspirin allergy or bleeding complications and patients |
| | 0. | unable or unwilling to tolerate anticoagulant/antiplatelet therapy and/or |
| | | non-responders to anticoagulant/antiplatelet therapy |
| | 9. | Fresh thrombus formation |
| | 10. | Patients with known hypersensitivity to the stent material (L605) and/or |
| | | PTFE |
| | 11. | The target lesion is either a modified TASC-II class C or D lesion with aortic |
| | | or common femoral lesion involvement: |
| | | <ul> <li>Type C lesions</li> <li>Unilateral External Iliac Artery stenosis</li> </ul> |
| | | <ul> <li>Unilateral External Iliac Artery stenosis<br/>extending into the Common Femoral Artery</li> </ul> |
| | | Unilateral External Iliac Artery occlusion that |
| | | involves the origins of the Internal Iliac and/or |
| | | Common Femoral Artery |
| | | Heavily calcified unilateral External Iliac Artery |
| | | occlusion with the involvement of the |
| | | Common Femoral Artery |
| | | <ul> <li>Type D lesions</li> </ul> |
| | | Infra-renal aortoiliac occlusion |
| | | Iliac stenoses in patients with an Abdominal Applie Applying (AAA), requiring tractments. |
| | | Aortic Aneurysm (AAA) requiring treatment |
| | | and not amenable to endograft placement or |

V2.00 dd20211119 2/4

<u>ID3 Medical - 20211119</u> BELSTREAM - Bard

| | other lesions requiring open aortic or iliac |
|---|---|
| | surgery |
| | Diffuse multiple stenoses involving the |
| | unilateral Common Iliac, External Iliac and |
| | Common Femoral Artery 12. Previously implanted stent(s) at the same lesion site |
| | Previously implanted stent(s) at the same lesion site |
| | 13. Reference segment diameter is not suitable for the available stent graft |
| | design |
| | 14. Untreatable lesion located at the distal outflow arteries |
| | 15. Use of alternative therapy (e.g. atherectomy, cutting balloon, DCB, laser, |
| | radiation therapy) as part of the index procedure |
| | 16. Patients refusing treatment |
| | 17. Patients for whom antiplatelet therapy, anticoagulants or thrombolytic |
| | drugs are contraindicated |
| | 18. Patients who exhibit persistent acute intraluminal thrombus of the |
| | proposed lesion site |
| | 19. Perforation at the angioplasty site evidenced by extravasation of contrast |
| | medium |
| | 20. Patients with a history of prior life-threatening contrast medium reaction |
| | 21. Patients with uncorrected bleeding disorders |
| | 22. Female patient with child bearing potential not taking adequate |
| | contraceptives or currently breastfeeding |
| | 23. Life expectancy of less than twelve months |
| | 24. Any planned surgical intervention/procedure within 30 days of the study |
| | procedure |
| | 25. Any patient considered to be hemodynamically unstable at onset of |
| | procedure |
| P.I. | Dr. Peter Goverde, ZNA Campus Stuivenberg, Antwerp, Belgium |
| Study conduct | The study will be conducted in accordance with the Declaration of Helsinki and ISO |
| | 14155:2011, and comply with requirements regarding Ethics Committees and any |
| | other applicable regulations |
| Participating sites | A.Z. Groeninge, Kortrijk, Belgium: Dr. Lerut |
| | A.Z. Sint-Blasius, Dendermonde, Belgium: Dr. Deloose |
| | Imelda Hospital, Bonheiden, Belgium: Dr. Verbist |
| | O.L.V. Hospital, Aalst, Belgium: Dr. Maene |
| | R.Z. H.H., Tienen, Belgium: Dr. Keirse |
| | Z.O.L., Genk, Belgium: Dr. Lansink |
| | Z.N.A. Stuivenberg, Antwerpen, Belgium: Dr. Goverde |
| • | · |

V2.00 dd20211119 3/4

<u>ID3 Medical - 20211119</u> <u>BELSTREAM - Bard</u>

Table 1. Study Investigations

| Time | | Tests and Procedures |
|-----------------------------------|----|-----------------------------------|
| Pre-Procedure | 1. | Medical History |
| (up to 24 hours before procedure, | 2. | Medication Registration |
| unless otherwise noted.) | 3. | Physical Exam |
| | 4. | Rutherford Categorization and ABI |
| Procedure | 1. | Angiography, pre–procedure |
| | 2. | Study inclusion |
| | 3. | Intervention |
| | 4. | Rutherford Categorization and ABI |
| One day Post-Procedure | 1. | Medication Registration |
| | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| One month Follow-up | 1. | Medication Registration |
| (± 7 days) | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| | 4. | Colour Flow Doppler Ultrasound |
| Six month Follow-up | 1. | Medication Registration |
| ( $\pm$ 30 days) | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| | 4. | Colour Flow Doppler Ultrasound |
| One year Follow-up | 1. | Medication Registration |
| ( $\pm$ 30 days) | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| | 4. | Colour Flow Doppler Ultrasound |
| Two year Follow-up | 1. | Medication Registration |
| (730 $\pm$ 30 days) | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| | 4. | Colour Flow Doppler Ultrasound |
| Three year Follow-up | 1. | Medication Registration |
| (1095 $\pm$ 30 days) | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| | 4. | Colour Flow Doppler Ultrasound |
| Four year Follow-up | 1. | Medication Registration |
| (1460 $\pm$ 30 days) | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| | 4. | Colour Flow Doppler Ultrasound |
| Five year Follow-up | 1. | Medication Registration |
| (1825 $\pm$ 30 days) | 2. | Physical Examination |
| | 3. | Rutherford Categorization and ABI |
| | 4. | Colour Flow Doppler Ultrasound |

## • Statistical Analysis Plan (SAP)

Descriptive data summaries will be used to present and summarize the collected data. For categorical variables (e.g. Gender) frequency distributions and cross tabulations will be given. For numeric variables (e.g. Patient age) minimum, maximum, mean, median and standard deviation will be calculated. For all variables a 95% confidence interval for the relevant parameters of the underlying distribution will be calculated. For all time-dependent events life-tables will be calculated using the Kaplan Meier estimate method, for a period starting on the date of the procedure up to and including the 60-month follow-up visit. Stratification to pre-procedural risk factors, Rutherford and lesion criteria will be performed and the log rank test will be used to compare between the different outcomes, associated p-values < 0.05 are defined as significant.

V2.00 dd20211119 4/4